CLINICAL TRIAL: NCT03114956
Title: Effects of Implant Surface Decontamination on Control of Peri-Implant Inflammation
Brief Title: Surface Decontamination in Treatment of Peri-Implantitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to secure funding
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Neema Bakhshalian, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-188
Record Dates: First submitted 2017-04-03; First posted 2017-04-14 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator who is analyzing the data will be blinded to the assigned groups to prevent bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Implant surface will be wiped with sterile gauze soaked alternatively in sterile saline and CHX (5 times)
  Interventions: Procedure: Gauze
- Group B (Experimental): Titanium brush: Titanium brush (TiBrush, Straumann, Switzerland) mounted on an oscillating hand piece will be used for 1 minute.
  Interventions: Procedure: Titanium brush
- Group C (Experimental): Air powder abrasion: One minute of air powder abrasion using Glycine prophy powder (Prophy Jet, Dentsply, USA) with overlapping passes form apical to coronal direction for 1 minute.
  Interventions: Procedure: Air powder abrasion
- Group D (Experimental): A comprehensive treatment including the use of titanium brush and air powder abrasion (as described above) and 30 seconds etching with 9.6% HF acid gel (Premier, USA) applied with a micro-applicator tip (Unipack Medical, USA), followed by copious irrigation with sterile saline.
  Interventions: Procedure: Comprehensive

INTERVENTIONS:
Procedure: Gauze — Implant surface will be wiped with sterile gauze soaked alternatively in sterile saline and CHX (5 times)
  Arms: Group A
Procedure: Titanium brush — Titanium brush: Titanium brush (TiBrush, Straumann, Switzerland) mounted on an oscillating hand piece will be used for 1 minute.
  Arms: Group B
Procedure: Air powder abrasion — Air powder abrasion: One minute of air powder abrasion using Glycine prophy powder (Prophy Jet, Dentsply, USA) with overlapping passes form apical to coronal direction for 1 minute.
  Arms: Group C
Procedure: Comprehensive — A comprehensive treatment including the use of titanium brush and air powder abrasion (as described above) and 30 seconds etching with 9.6% HF acid gel (Premier, USA) applied with a micro-applicator tip (Unipack Medical, USA), followed by copious irrigation with sterile saline.
  Arms: Group D

SUMMARY:
Peri-implantitis represents a major biological complication of implant dentistry with reported prevalence of up to 47% of implants. The disease is characterized by inflammatory response to the biofilm inhabiting the implant surface. To treat this inflammatory disease, surgical and non-surgical therapies have been proposed, all of which entail biofilm removal through implant surface decontamination. Systematic review of various surface decontamination protocols has failed to demonstrate superiority of any of the protocols. One possible explanation is that most studies have examined decontamination of implant surfaces following experimentally-induced peri-implantitis, where implant surfaces lack the tenacious mineralized biofilm often found in clinical peri-implantitis and are therefore easily decontaminated.

The investigators have hypothesized that control of inflammation and repair of pathologically damaged peri-implant tissues requires a comprehensive mechanical plus chemical surface decontamination therapy. The aims of this study are to 1) determine the most effective surface decontamination protocol that can lead to control of peri-implant inflammation and 2) delineate the microbial and immunological mediators that are associated with the changes in peri-implant inflammation. The investigators propose to compare conventional implant surface contamination techniques to a comprehensive mechanical plus chemical protocol. This randomized controlled clinical trial seeks to enroll 68 participants with at least one implant diagnosed with moderate to severe peri-implantitis. Pre-op parameters to be assessed include: probing pocket depth, bleeding on probing, suppuration, plaque index, marginal inflammation, recession, clinical attachment level, inflammatory biomarkers and microbial sampling, and digital intra-oral peri-apical radiograph. Subjects will be randomly assigned to one of the four surgical debridement intervention groups: (A) gauzes soaked in sterile saline and chlorhexidine; (B) Titanium brush; (C) Air power abrasion; (D) comprehensive surface decontamination, including titanium brush, air powder abrasion and surface etching with 9.6% hydrofluoric acid gel. At 3-months post-operative, the initial clinical assessment will be repeated. The clinical examination will be used to analyze the efficacy of each treatment in controlling peri-implant mucosal inflammation. The ultimate objective of this research is not only to identify an effective method for control of peri-implant inflammation, but also to lay the foundation to detect biomarkers of peri-implantitis that can potentially be helpful in future studies as risk factors of this disease.

ELIGIBILITY:
Inclusion Criteria:

* PPD >6 mm
* Positive BOP
* Peri-implant marginal bone loss (MBL) >3 mm
* Age: 18 to 75 years

Exclusion Criteria

* Implant mobility
* Smoking
* Current cancer
* Steroids use (last 2 years)
* Bisphosphonates use (last 4 years)
* Uncontrolled diabetes (HBA1c >7)
* Other systemic conditions that affect wound healing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Bleeding on Probing (BOP) | 3 months
  A periodontal probe will be used at 6 locations around each implant (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, and distolingual). Presence of gingival bleeding upon probing will be recorded. This will be a binary outcome (Yes or No)
Suppuration upon probing | 3 months
  A periodontal probe will be used at 6 locations around each implant (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, and distolingual). Presence of suppuration upon probing will be recorded. This will be a binary outcome (Yes or No)
Probing Pocket Depth (PPD) | 3 months
  Distance from the gingival margin to the depth of the pocket

SECONDARY OUTCOMES:
Marginal bone loss | 3 month
  Measurement from the implant platform to first bone-to-implant contact
Inflammatory biomarkers | 3 months
  Inflammatory biomarkers in the peri-implant crevicular fluid (PICF)
Microbial profile | 3 months
  Microbial profile in the peri-implant crevicular fluid (PICF)

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, the clinical data and radiographs will be shared with other investigators included in this study for analysis.